CLINICAL TRIAL: NCT00464945
Title: A Phase 3, Randomised,Active-Controlled ,Double-Blind Trial Evaluating the Safety, Tolerability, and Immunogenicity of Manufacturing Scale 13-valent Pneumococcal Conjugate Vaccine
Brief Title: Wyeth Study To Evaluate a 13-valent Pneumococcal Conjugate Vaccine in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6096A1-3000
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Results first posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-07

CONDITIONS: Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- 2 (Active Comparator)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine — 1 dose at 2,3,4 and 12 months of age

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of manufacturing scale 13-valent pneumococcal conjugate (13vPnC) vaccine compared to pilot scale 13vPnC in healthy infants when given with routine pediatric vaccines.

ELIGIBILITY:
Inclusion criteria:

1. Aged 2 months (42 to 98 days) at time of enrollment.
2. Available for entire study period and whose parent/legal guardian can be reached by telephone.
3. Healthy infant as determined by medical history, physical examination, and judgment of the investigator.
4. Parent/legal guardian must be able to complete all relevant study procedures during study participation.

Exclusion criteria:

1. Previous vaccination with licensed or investigational pneumococcal, Hib conjugate, diphtheria, tetanus, pertussis, or polio vaccines.
2. A previous anaphylactic reaction to any vaccine or vaccine-related component.
3. Contraindication to vaccination with Hib conjugate, diphtheria, tetanus, pertussis, polio, hepatitis B, measles, mumps, rubella, or pneumococcal vaccines.
4. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
5. Known or suspected immune deficiency or suppression.
6. History of culture-proven invasive disease caused by S pneumoniae.
7. Major known congenital malformation or serious chronic disorders.
8. Significant neurological disorder or history of seizure including febrile seizure, or significant stable or evolving disorders such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorders. Does not include resolving syndromes due to birth trauma such as Erb palsy.
9. Receipt of blood products or gamma-globulin (including hepatitis B immunoglobulin and monoclonal antibodies; eg, Synagis®).
10. Participation in another investigational or interventional trial. Participation in purely observational studies is acceptable.
11. Infant who is a direct descendant (child or grandchild) of a member of the study site personnel.

Ages: 41 Days to 99 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 269 (Actual)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com
Locations (7):
- Poland (7):
  - Torun, Bydgoszcz
  - Krakow, Krakow
  - Siemianowice Śląskie, Krakow
  - Lubartowie, Lublin Voivodeship
  - Lublin, Lublin Voivodeship
  - Warsaw, Warszawa
  - Lodz, Łódź Voivodeship

REFERENCES:
- [Derived] Gadzinowski J, Albrecht P, Hasiec B, Konior R, Dziduch J, Witor A, Mellelieu T, Tansey SP, Jones T, Sarkozy D, Emini EA, Gruber WC, Scott DA. Phase 3 trial evaluating the immunogenicity, safety, and tolerability of manufacturing scale 13-valent pneumococcal conjugate vaccine. Vaccine. 2011 Apr 5;29(16):2947-55. doi: 10.1016/j.vaccine.2011.02.002. Epub 2011 Feb 16. PMID 21335032

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Poland from June 2007 to August 2007.
Pre-assignment Details: Participants were enrolled into the study according to inclusion/exclusion criteria without a screening period.
Groups:
- 13vPnC Manufacturing: Participants received one single 0.5mL manufacturing scale dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined diphtheria, tetanus, and acellular pertussis inactivated poliovirus, and hemophilus influenza type b vaccine (DTaP-IPV-Hib) and hepatitis B virus vaccine (HBV) at 2 months (infant series, dose 1). Participants received one single 0.5mL manufacturing scale dose of 13vPnC coadministered with DTaP-IPV-Hib at 3 and 4 months (infant series, dose 2 and 3). Participants received one single 0.5mL manufacturing scale dose of 13vPnC coadministered with measles, mumps, and rubella vaccine (MMR) and 12 months of age (toddler dose).
- 13vPnC Pilot: Participants received one single 0.5mL pilot scale dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined diphtheria, tetanus, and acellular pertussis inactivated poliovirus, and hemophilus influenza type b vaccine (DTaP-IPV-Hib) and hepatitis B virus vaccine (HBV) at 2 months (infant series, dose 1). Participants received one single 0.5mL pilot scale dose of 13vPnC coadministered with DTaP-IPV-Hib at 3 and 4 months (infant series, dose 2 and 3). Participants received one single 0.5mL pilot scale dose of 13vPnC coadministered with measles, mumps, and rubella vaccine (MMR) and 12 months of age (toddler dose).
Period: Infant Series
Arm/Group | 13vPnC Manufacturing | 13vPnC Pilot
Started | 135 | 134
Vaccinated Dose 1 | 134 | 134
Vaccinated Dose 2 | 132 | 133
Vaccinated Dose 3 | 132 | 133
Completed | 131 | 133
Not Completed | 4 | 1
Not completed — Withdrawal by parent/guardian request | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: After Infant Series
Arm/Group | 13vPnC Manufacturing | 13vPnC Pilot
Started | 131 | 133
Completed | 131 | 131
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Toddler Dose
Arm/Group | 13vPnC Manufacturing | 13vPnC Pilot
Started | 131 | 131
Completed | 131 | 130
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC Manufacturing | 13vPnC Pilot | Total
Number analyzed (Participants) | 135 | 134 | 269
Age Continuous [Mean (Standard Deviation); unit: months] | 2.1 (0.6) | 2.1 (0.5) | 2.1 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 67 | 132
  Male | 70 | 67 | 137

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Antibody Level ≥0.35μg/mL in 13vPnC Manufacturing Scale Group Relative to 13vPnC Pilot Scale Group After the 3-Dose Infant Series
Description: Percentages of participants achieving WHO predefined antibody threshold ≥0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after 3-dose infant series (5 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Manufacturing | 13vPnC Pilot
Number analyzed (Participants) | 128 | 131
percentage of participants
  Common Serotypes-Serotype 4 | 97.7 [93.3 to 99.5] | 96.9 [92.4 to 99.2]
  Common Serotypes-Serotype 6B | 77.3 [69.1 to 84.3] | 74.0 [65.7 to 81.3]
  Common Serotypes-Serotype 9V | 98.4 [94.5 to 99.8] | 96.2 [91.3 to 98.7]
  Common Serotypes-Serotype 14 | 92.9 [87.0 to 96.7] | 94.5 [89.1 to 97.8]
  Common Serotypes-Serotype 18C | 96.1 [91.1 to 98.7] | 93.1 [87.4 to 96.8]
  Common Serotypes-Serotype 19F | 98.4 [94.4 to 99.8] | 97.7 [93.5 to 99.5]
  Common Serotypes-Serotype 23F | 82.8 [75.1 to 88.9] | 81.7 [74.0 to 87.9]
  Additional Serotypes-Serotype 1 | 93.0 [87.1 to 96.7] | 90.8 [84.5 to 95.2]
  Additional Serotypes-Serotype 3 | 93.7 [88.0 to 97.2] | 95.4 [90.3 to 98.3]
  Additional Serotypes-Serotype 5 | 90.6 [84.2 to 95.1] | 88.5 [81.8 to 93.4]
  Additional Serotypes-Serotype 6A | 85.2 [77.8 to 90.8] | 86.3 [79.2 to 91.6]
  Additional Serotypes-Serotype 7F | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]
  Additional Serotypes-Serotype 19A | 99.2 [95.7 to 100.0] | 99.2 [95.8 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 4 the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = 0.7, 95% CI [-3.9 to 5.6]
Statistical Analysis 2: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 6B the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = 3.3, 95% CI [-7.3 to 13.8]
Statistical Analysis 3: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 9V the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = 2.3, 95% CI [-2.1 to 7.3]
Statistical Analysis 4: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 14 the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = -1.6, 95% CI [-8.2 to 4.7]
Statistical Analysis 5: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 18C the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = 3.0, 95% CI [-2.8 to 9.2]
Statistical Analysis 6: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 19F the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = 0.7, 95% CI [-3.5 to 5.1]
Statistical Analysis 7: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 23F the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = 1.1, 95% CI [-8.4 to 10.6]
Statistical Analysis 8: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 1 the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = 2.1, 95% CI [-4.8 to 9.2]
Statistical Analysis 9: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 3 the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = -1.7, 95% CI [-7.9 to 4.2]
Statistical Analysis 10: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 5 the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = 2.1, 95% CI [-5.6 to 9.9]
Statistical Analysis 11: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 6A the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = -1.1, 95% CI [-9.9 to 7.6]
Statistical Analysis 12: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 7F the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = 0.0, 95% CI [-3.0 to 2.8]
Statistical Analysis 13: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 19A the difference in percentages between the two groups (13vPnC Manufacturing - 13vPnC Pilot) was calculated; Test type: Superiority or Other; Difference = -0.0, 95% CI [-3.6 to 3.5]

2. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant(Sig) (present and interfered with limb movement). Induration and erythema were scaled as Any (induration or erythema present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (Mod) (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all participants who received at least 1 dose of vaccine; (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC Manufacturing Dose 1: Participants received one single 0.5mL manufacturing scale dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined diphtheria, tetanus, and acellular pertussis inactivated poliovirus, and hemophilus influenza type b vaccine (DTaP-IPV-Hib) and hepatitis B virus vaccine (HBV) at 2 months (infant series, dose 1).
- 13vPnC Pilot Dose 1: Participants received one single 0.5mL pilot scale dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined diphtheria, tetanus, and acellular pertussis inactivated poliovirus, and hemophilus influenza type b vaccine (DTaP-IPV-Hib) and hepatitis B virus vaccine (HBV) at 2 months (infant series, dose 1).
- 13vPnC Manufacturing Dose 2; 13vPnC Manufacturing Dose 3: Participants received one single 0.5mL manufacturing scale dose of 13vPnC coadministered with DTaP-IPV-Hib at 3 and 4 months (infant series, dose 2 and 3).
- 13vPnC Pilot Dose 2; 13vPnC Pilot Dose 3: Participants received one single 0.5mL pilot scale dose of 13vPnC coadministered with DTaP-IPV-Hib at 3 and 4 months (infant series, dose 2 and 3).
- 13vPnC Manufacturing Toddler Dose: Participants received one single 0.5mL manufacturing scale dose of 13vPnC coadministered with measles, mumps, and rubella vaccine (MMR) and 12 months of age (toddler dose).
- 13vPnC Pilot Toddler Dose: Participants received one single 0.5mL pilot scale dose of 13vPnC coadministered with measles, mumps, and rubella vaccine (MMR) and 12 months of age (toddler dose).
Arm/Group | 13vPnC Manufacturing Dose 1 | 13vPnC Pilot Dose 1 | 13vPnC Manufacturing Dose 2 | 13vPnC Pilot Dose 2 | 13vPnC Manufacturing Dose 3 | 13vPnC Pilot Dose 3 | 13vPnC Manufacturing Toddler Dose | 13vPnC Pilot Toddler Dose
Number analyzed (Participants) | 134 | 134 | 132 | 133 | 132 | 133 | 131 | 131
percentage of participants
  Tenderness-Any (n=133,130,128,128,124,119,115,117) | 18.8 | 20.0 | 20.3 | 17.2 | 15.3 | 12.6 | 24.3 | 29.1
  Tenderness-Sig (n=131,129,128,128,124,119,112,114) | 0.8 | 3.9 | 1.6 | 3.1 | 1.6 | 0.0 | 1.8 | 3.5
  Swelling-Any (n=132,130,129,129,126,122,113,115) | 25.0 | 20.0 | 30.2 | 27.1 | 29.4 | 30.3 | 22.1 | 26.1
  Swelling-Mild (n=132,130,129,129,126,121,113,115) | 22.7 | 17.7 | 29.5 | 25.6 | 27.0 | 25.6 | 22.1 | 25.2
  Swelling-Mod (n=132,129,128,128,124,120,113,114) | 6.1 | 7.0 | 8.6 | 8.6 | 8.9 | 13.3 | 8.8 | 8.8
  Swelling-Severe(n=131,129,128,128,124,119,112,113) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Redness-Any (n=132,131,129,131,125,123,115,116) | 28.8 | 24.4 | 37.2 | 33.6 | 40.0 | 34.1 | 37.4 | 42.2
  Redness-Mild (n=132,131,129,131,125,123,115,115) | 28.8 | 22.9 | 36.4 | 33.6 | 38.4 | 33.3 | 33.9 | 36.5
  Redness-Mod (n=131,129,128,128,124,119,113,114) | 0.0 | 1.6 | 3.1 | 1.6 | 5.6 | 3.4 | 10.6 | 12.3
  Redness-Severe(n=131,129,128,128,124,119,112,113) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.9

3. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events (Infant Series)
Description: Systemic events (fever ≥ 38 degrees Celsius [C] but ≤ 39 C, fever >39 C but ≤ 40 C, fever > 40 C, decreased appetite, irritability, increased sleep, decreased sleep, use of medication (Meds)to prevent symptoms (sx), and use of medication to treat symptoms) were collected using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all participants (268) who received at least 1 dose of vaccine; (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Manufacturing Dose 1 | 13vPnC Pilot Dose 1 | 13vPnC Manufacturing Dose 2 | 13vPnC Pilot Dose 2 | 13vPnC Manufacturing Dose 3 | 13vPnC Pilot Dose 3
Number analyzed (Participants) | 134 | 134 | 132 | 133 | 132 | 133
percentage of participants
  Fever ≥38°C but ≤39°C (n=132,130,129,130,124,121) | 18.2 | 19.2 | 16.3 | 20.0 | 11.3 | 17.4
  Fever >39°C but ≤40°C (n=131,129,128,128,124,119) | 0.8 | 0.8 | 0.8 | 1.6 | 0.0 | 3.4
  Fever >40°C (n=131,129,128,128,124,119) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Decreased appetite (n=133,129,129,128,125,121) | 20.3 | 24.0 | 14.7 | 15.6 | 16.8 | 19.0
  Irritability (n=134,131,130,131,127,123) | 50.0 | 51.9 | 53.8 | 49.6 | 41.7 | 37.4
  Increased sleep (n=132,129,128,129124,121) | 41.7 | 39.5 | 25.0 | 29.5 | 20.2 | 30.6
  Decreased sleep (n=132,130,129,129,124,123) | 27.3 | 32.3 | 24.0 | 20.9 | 18.5 | 19.5
  Meds to treat sx (n=132,130,128,128,124,123) | 12.9 | 17.7 | 13.3 | 14.1 | 8.9 | 14.6
  Meds to prevent sx (n=132,130,128,129124,121) | 12.9 | 9.2 | 11.7 | 10.1 | 10.5 | 8.3

4. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events (Toddler Series)
Description: Systemic events (fever ≥ 38 degrees Celsius [C] but ≤ 39 C, fever >39 C but ≤ 40 C, fever > 40 C), decreased appetite, irritability, increased sleep, decreased sleep, use of medication to prevent symptoms, and use of medication to treat symptoms) were collected using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after toddler dose
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC Manufacturing: Participants received one single 0.5mL manufacturing scale dose of 13vPnC coadministered with measles, mumps, and rubella vaccine (MMR) and 12 months of age (toddler dose).
- 13vPnC Pilot: Participants received one single 0.5mL pilot scale dose of 13vPnC coadministered with measles, mumps, and rubella vaccine (MMR) and 12 months of age (toddler dose).
Arm/Group | 13vPnC Manufacturing | 13vPnC Pilot
Number analyzed (Participants) | 131 | 131
percentage of participants
  Fever ≥38°C but ≤39°C (n=114,114) | 14.0 | 13.2
  Fever >39°C but ≤40°C (n=112,113) | 0.9 | 0.9
  Fever >40°C (n=112,113) | 0.0 | 0.0
  Decreased appetite (n=115,117) | 20.9 | 23.1
  Irritability (n=119,123) | 40.3 | 44.7
  Increased sleep (n=114,119) | 18.4 | 16.8
  Decreased sleep (n=116,117) | 13.8 | 13.7
  Medication to treat symptoms (n=113,115) | 17.7 | 17.4
  Medication to prevent symptoms (n=114,114) | 12.3 | 12.3

5. Primary Outcome: Geometric Mean Antibody Concentration in 13vPnC Manufacturing Scale Group Relative to 13vPnC Pilot Scale Group After the 3-Dose Infant Series
Description: Antibody concentration/geometric mean concentration (GMC) as measured by enzyme-linked immunosorbent assay (ELISA) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after 3-dose infant series (5 months of age)
Population: Evaluable immunogenicity (per protocol) population were participants who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- 13vPnC Manufacturing: Participants received one single 0.5mL manufacturing scale dose of 13vPnC coadministered with Infanrix hexa at 2, 3, 4 months (infant series) and 12 months of age (toddler dose).
- 13vPnC Pilot: Participants received one single 0.5mL pilot scale dose of 13vPnC coadministered with Infanrix hexa at 2, 3, 4 months (infant series) and 12 months of age (toddler dose).
Arm/Group | 13vPnC Manufacturing | 13vPnC Pilot
Number analyzed (Participants) | 128 | 131
μg/mL
  Common Serotypes-Serotype 4 | 2.09 [1.81 to 2.40] | 1.55 [1.34 to 1.79]
  Common Serotypes - Serotype 6B | 0.80 [0.65 to 0.98] | 0.83 [0.66 to 1.06]
  Common Serotypes - Serotype 9V | 1.28 [1.13 to 1.43] | 1.21 [1.08 to 1.37]
  Common Serotypes - Serotype 14 | 2.15 [1.77 to 2.61] | 2.30 [1.91 to 2.77]
  Common Serotypes - Serotype 18C | 1.60 [1.38 to 1.87] | 1.51 [1.31 to 1.75]
  Common Serotypes - Serotype 19F | 1.60 [1.40 to 1.83] | 1.64 [1.44 to 1.86]
  Common Serotypes - Serotype 23F | 0.82 [0.69 to 0.98] | 0.92 [0.77 to 1.10]
  Additional Serotypes - Serotype 1 | 1.42 [1.21 to 1.66] | 1.29 [1.10 to 1.51]
  Additional Serotypes - Serotype 3 | 1.20 [1.05 to 1.38] | 1.21 [1.06 to 1.37]
  Additional Serotypes - Serotype 5 | 0.96 [0.84 to 1.09] | 1.00 [0.87 to 1.16]
  Additional Serotypes - Serotype 6A | 0.87 [0.74 to 1.03] | 1.05 [0.89 to 1.25]
  Additional Serotypes - Serotype 7F | 2.00 [1.77 to 2.25] | 2.14 [1.89 to 2.42]
  Additional Serotypes - Serotype 19A | 2.19 [1.91 to 2.50] | 2.31 [2.05 to 2.61]
Statistical Analysis 1: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 4 the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 1.35, 95% CI [1.10 to 1.65]
Statistical Analysis 2: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 6B the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 0.96, 95% CI [0.70 to 1.31]
Statistical Analysis 3: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 9V the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 1.05, 95% CI [0.89 to 1.24]
Statistical Analysis 4: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 14 the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 0.93, 95% CI [0.71 to 1.22]
Statistical Analysis 5: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 18C the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 1.06, 95% CI [0.86 to 1.30]
Statistical Analysis 6: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 19F the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 0.98, 95% CI [0.81 to 1.17]
Statistical Analysis 7: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 23F the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 0.90, 95% CI [0.70 to 1.15]
Statistical Analysis 8: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 1 the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 1.10, 95% CI [0.88 to 1.37]
Statistical Analysis 9: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 3 the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 1.00, 95% CI [0.83 to 1.20]
Statistical Analysis 10: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 5 the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 0.95, 95% CI [0.79 to 1.16]
Statistical Analysis 11: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 6A the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 0.83, 95% CI [0.66 to 1.05]
Statistical Analysis 12: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 7F the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 0.93, 95% CI [0.79 to 1.11]
Statistical Analysis 13: Comparison: 13vPnC Manufacturing vs 13vPnC Pilot; For serotype 19A the GMC ratio was calculated; Test type: Superiority or Other; Ratio = 0.95, 95% CI [0.79 to 1.13]

ADVERSE EVENTS:
Groups:
- 13vPnC Manufacturing Infant Series: Participants received one single 0.5mL manufacturing scale dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined diphtheria, tetanus, and acellular pertussis inactivated poliovirus, and hemophilus influenza type b vaccine (DTaP-IPV-Hib) and hepatitis B virus vaccine (HBV) at 2 months (infant series, dose 1). Participants received one single 0.5mL manufacturing scale dose of 13vPnC coadministered with DTaP-IPV-Hib at 3 and 4 months (infant series, dose 2 and 3).
- 13vPnC Pilot Infant Series: Participants received one single 0.5mL pilot scale dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined diphtheria, tetanus, and acellular pertussis inactivated poliovirus, and hemophilus influenza type b vaccine (DTaP-IPV-Hib) and hepatitis B virus vaccine (HBV) at 2 months (infant series, dose 1). Participants received one single 0.5mL pilot scale dose of 13vPnC coadministered with DTaP-IPV-Hib at 3 and 4 months (infant series, dose 2 and 3).
- 13vPnC Manufacturing Post-Infant Series: Participants received one single 0.5mL manufacturing scale dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined diphtheria, tetanus, and acellular pertussis inactivated poliovirus, and hemophilus influenza type b vaccine (DTaP-IPV-Hib) and hepatitis B virus vaccine (HBV) at 2 months (infant series, dose 1). Participants received one single 0.5mL manufacturing scale dose of 13vPnC coadministered with DTaP-IPV-Hib at 3 and 4 months (infant series, dose 2 and 3). Assessment done at 5 months of age, 1 month after infant series.
- 13vPnC Pilot Post-Infant Series: Participants received one single 0.5mL pilot scale dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined diphtheria, tetanus, and acellular pertussis inactivated poliovirus, and hemophilus influenza type b vaccine (DTaP-IPV-Hib) and hepatitis B virus vaccine (HBV) at 2 months (infant series, dose 1). Participants received one single 0.5mL pilot scale dose of 13vPnC coadministered with DTaP-IPV-Hib at 3 and 4 months (infant series, dose 2 and 3). Assessment done at 5 months of age, 1 month after infant series.
- 13vPnC Manufacturing Toddler Series: Participants received one single 0.5mL manufacturing scale dose of 13vPnC coadministered with measles, mumps, and rubella vaccine (MMR) and 12 months of age (toddler dose).
- 13vPnC Pilot Toddler Series: Participants received one single 0.5mL pilot scale dose of 13vPnC coadministered with measles, mumps, and rubella vaccine (MMR) and 12 months of age (toddler dose).
Arm/Group | 13vPnC Manufacturing Infant Series | 13vPnC Pilot Infant Series | 13vPnC Manufacturing Post-Infant Series | 13vPnC Pilot Post-Infant Series | 13vPnC Manufacturing Toddler Series | 13vPnC Pilot Toddler Series
Serious Adverse Events (participants affected / at risk) | 4/134 | 2/134 | 10/134 | 11/134 | 0/131 | 1/131
Other Adverse Events (participants affected / at risk) | 70/134 | 68/134 | 3/134 | 7/134 | 48/131 | 55/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Manufacturing Infant Series (N=134) | 13vPnC Pilot Infant Series (N=134) | 13vPnC Manufacturing Post-Infant Series (N=134) | 13vPnC Pilot Post-Infant Series (N=134) | 13vPnC Manufacturing Toddler Series (N=131) | 13vPnC Pilot Toddler Series (N=131)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 2 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Crying (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 3 | 4 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 3 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Manufacturing Infant Series (N=134) | 13vPnC Pilot Infant Series (N=134) | 13vPnC Manufacturing Post-Infant Series (N=134) | 13vPnC Pilot Post-Infant Series (N=134) | 13vPnC Manufacturing Toddler Series (N=131) | 13vPnC Pilot Toddler Series (N=131)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 2 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hip dysplasia (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Plagiocephaly (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 5 | 4 | 0 | 0 | 1 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 0 | 0 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Enlarged uvula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 2 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Milk allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 12 | 10 | 0 | 0 | 1 | 2
Pharyngitis (Infections and infestations) | 9 | 10 | 0 | 0 | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 8 | 11 | 0 | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 8 | 9 | 0 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 5 | 7 | 0 | 0 | 1 | 2
Candidiasis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 3
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Rickets (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Crying (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Psychomotor retardation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Posthitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 25/133 | 26/130 | 0 | 0 | 28/115 | 34/117 — Dose 1 Infant Series and Toddler Dose
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 26/128 | 22/128 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 19/124 | 15/119 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 1/131 | 5/129 | 0 | 0 | 2/112 | 4/114 — Dose 1 Infant Series and Toddler Dose
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 2/128 | 4/128 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 2/124 | 0/119 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Induration (Any) (Skin and subcutaneous tissue disorders) | 33/132 | 26/130 | 0 | 0 | 25/113 | 30/115 — Dose 1 Infant Series and Toddler Dose
Induration (Any) (Skin and subcutaneous tissue disorders) | 39/129 | 35/129 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Induration (Any) (Skin and subcutaneous tissue disorders) | 37/126 | 37/122 | 0 | 0 | 0 | 0 — Dose 3 Infant Serie
Induration (Mild) (Skin and subcutaneous tissue disorders) | 30/132 | 23/130 | 0 | 0 | 25/113 | 29/115 — Dose 1 Infant Series and Toddler Dose
Induration (Mild) (Skin and subcutaneous tissue disorders) | 38/129 | 33/129 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Induration(Mild) (Skin and subcutaneous tissue disorders) | 34/126 | 31/121 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 8/132 | 9/129 | 0 | 0 | 10/113 | 10/114 — Dose 1 Infant Series and Toddler Dose
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 11/128 | 11/128 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 11/124 | 16/120 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/131 | 0/129 | 0 | 0 | 0/112 | 0/113 — Dose 1 Infant Series and Toddler Dose
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/128 | 0/128 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/124 | 0/119 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Erythema (Any) (Skin and subcutaneous tissue disorders) | 38/132 | 32/131 | 0 | 0 | 43/115 | 49/116 — Dose 1 Infant Series and Toddler Dose
Erythema (Any) (Skin and subcutaneous tissue disorders) | 48/129 | 44/131 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Erythema (Any) (Skin and subcutaneous tissue disorders) | 50/125 | 42/123 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 38/132 | 30/131 | 0 | 0 | 39/115 | 42/115 — Dose 1 Infant Series and Toddler Dose
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 47/129 | 44/131 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 48/125 | 41/123 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 0/131 | 2/129 | 0 | 0 | 12/113 | 14/114 — Dose 1 Infant Series and Toddler Dose
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 4/128 | 2/128 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 7/124 | 4/119 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/131 | 0/129 | 0 | 0 | 0/112 | 1/113 — Dose 1 Infant Series and Toddler Dose
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/128 | 0/128 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/124 | 0/119 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Fever ≥38°C but ≤39°C (General disorders) | 24/132 | 25/130 | 0 | 0 | 16/114 | 15/114 — Dose 1 Infant Series and Toddler Dose
Fever ≥38°C but ≤39°C (General disorders) | 21/129 | 26/130 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Fever ≥38°C but ≤39°C (General disorders) | 14/124 | 21/121 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Fever >39°C but ≤40°C (General disorders) | 1/131 | 1/129 | 0 | 0 | 1/112 | 1/113 — Dose 1 Infant Series and Toddler Dose
Fever >39°C but ≤40°C (General disorders) | 1/128 | 2/128 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Fever >39°C but ≤40°C (General disorders) | 0/124 | 4/119 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Fever >40°C (General disorders) | 0/131 | 0/129 | 0 | 0 | 0/112 | 0/113 — Dose 1 Infant Series and Toddler Dose
Fever >40°C (General disorders) | 0/128 | 0/128 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Fever >40°C (General disorders) | 0/124 | 0/119 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Decreased appetite (General disorders) | 27/133 | 31/129 | 0 | 0 | 24/115 | 27/117 — Dose 1 Infant Series and Toddler Dose
Decreased appetite (General disorders) | 19/129 | 20/128 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Decreased appetite (General disorders) | 21/125 | 23/121 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Irritability (General disorders) | 67 | 68/131 | 0 | 0 | 48/119 | 55/123 — Dose 1 Infant Series and Toddler Dose
Irritability (General disorders) | 70/130 | 65/131 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Irritability (General disorders) | 53/127 | 46/123 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Increased sleep (General disorders) | 55/132 | 51/129 | 0 | 0 | 21/114 | 20/119 — Dose 1 Infant Series and Toddler Dose
Increased sleep (General disorders) | 32/128 | 38/129 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Increased sleep (General disorders) | 25/124 | 37/121 | 0 | 0 | 0 | 0 — Dose 3 Infant Series
Decreased sleep (General disorders) | 36/132 | 42/130 | 0 | 0 | 16/116 | 16/117 — Dose 1 Infant Series and Toddler Dose
Decreased sleep (General disorders) | 31/129 | 27/129 | 0 | 0 | 0 | 0 — Dose 2 Infant Series
Decreased sleep (General disorders) | 23/124 | 24/123 | 0 | 0 | 0 | 0 — Dose 3 Infant Series

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.